CLINICAL TRIAL: NCT03557294
Title: Varenicline OTC Trial on Efficacy and Safety
Acronym: VOTC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Los Angeles Clinical Trials (Unknown); University of Nevada, Reno (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DA044125 (NIH); R01DA044125 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-06-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Dependence; Withdrawal Symptoms; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Substance Withdrawal Syndrome; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1.0mg varenicline b.i.d. (Experimental): Days 1 through 3: 0.5mg, once daily; days 4 through 7: 0.5mg, twice daily; days 8 through end of treatment: 1mg, twice daily.
  Interventions: Drug: 1.0mg Varenicline b.i.d.
- 0.5mg varenicline b.i.d. (Experimental): Days 1 through 3: 0.5mg, once daily; 0.5 mg b.i.d. dose starting at day 4 through the end of the study
  Interventions: Drug: 0.5mg Varenicline b.i.d.
- 0.0mg placebo varenicline b.i.d. (Placebo Comparator): Days 1 through 3: 0.0mg placebo once daily; days 4 through 7: 0.0mg placebo twice daily; days 8 through end of treatment: 0.0 mg placebo twice daily.
  Interventions: Drug: 0.0mg placebo Varenicline b.i.d.

INTERVENTIONS:
Drug: 1.0mg Varenicline b.i.d. — Varenicline is classified as a selective nicotine receptor partial agonist (SNRPA) that works both to stimulate the nicotine receptor and block smoking reward at the α4β2 nicotinic receptor subtype.
  Arms: 1.0mg varenicline b.i.d.
Drug: 0.5mg Varenicline b.i.d. — Varenicline is classified as a selective nicotine receptor partial agonist (SNRPA) that works both to stimulate the nicotine receptor and block smoking reward at the α4β2 nicotinic receptor subtype.
  Arms: 0.5mg varenicline b.i.d.
Drug: 0.0mg placebo Varenicline b.i.d. — Product that looks like active varenicline, but contains no active ingredient
  Arms: 0.0mg placebo varenicline b.i.d.

SUMMARY:
The primary goal of the proposed research is to test whether varenicline (Chantix) is safe and effective as an over-the-counter (OTC) medication.

DETAILED DESCRIPTION:
Given the recent research on varenicline showing that it is more effective than nicotine patch and bupropion, and with the removal of the box warning, research is needed to assess whether smokers can use varenicline without a prescription and formal behavioral support. To test this, the primary goal of the proposed research is to test whether varenicline is a candidate for switching from prescription (Rx) to OTC, and whether a dose lower than that currently approved is as effective in an OTC environment. To understand the within-person mechanisms explaining how and when OTC varenicline might improve cessation outcomes, the investigators also propose to assess experience with OTC varenicline via (a) ecological momentary assessment (EMA).

Primary Objectives:

1. To assess the safety and effectiveness of the current FDA-approved 1 mg b.i.d. varenicline for smoking cessation in comparison with placebo when used in a simulated OTC study condition.
2. To assess the safety and effectiveness of .5mg b.i.d. varenicline in comparison with 1mg b.i.d. varenicline and placebo when used in a simulated OTC study condition.

ELIGIBILITY:
Inclusion Criteria for the In-person Cohort

1. 21 years of age or older
2. Self-reported daily smoker
3. Breath CO > 10ppm
4. Motivated to quit smoking completely within five weeks of the Screening Visit (>5 on reported motivation)
5. Capable of and agree to complete study requirements
6. Literate in English, self-report
7. Must be available for the duration of study
8. Informed consent obtained
9. Willing and able to provide additional data between visits using ecological momentary assessment (EMA)
10. Must own study compatible smart-phone (iPhone or Android)

Exclusion Criteria for the In-person Cohort

1. Any self-report, diagnosis or treatment of heart attack, unstable angina, angioedema, seizures, cerebrovascular accident (CVA) within the last six months.
2. Any self-report, diagnosis or treatment of bipolar, schizophrenia or suicidal ideation within the last six months. (For suicidal ideation a score of ≥7 on the Suicidal Behavior Questionnaire, see Appendix 15)
3. Self-report of diagnosis or treatment for depression within the past six months, unless participant has written permission by their healthcare provider to participate
4. Systolic blood pressure 160 or higher and/or diastolic blood pressure 100 or higher (see site applicable SOP for Evaluating and Reporting Blood Pressure and Appendices 5 and 6 for participant handouts)
5. History of renal disease
6. Allergy to any of the ingredients in varenicline
7. Participation in another smoking cessation program or any type of clinical trial in the past 3 months
8. Use of any smoking cessation medication in the past three months
9. Any other medical condition(s) which the licensed study physician deems unacceptable for participation in this study
10. Positive drug screen indicating possible substance abuse (eg opiates, amphetamines, benzodiazepines, cocaine or other substances), unless participant can show that the medication has been prescribed by licensed clinical provider.
11. Consume greater than 21 alcohol drinks per week.
12. No two members of the same household may participate in this study
13. No study staff or their immediate family may participate in the study
14. Females who are pregnant, breast feeding, or not currently using a medically approved form of birth control and unwilling to do so.

Acceptable methods of birth control include abstinence, oral contraceptives, the contraceptive patch, the contraceptive ring, and condoms.

Inclusion Criteria for the Remote Cohort

1. 21 years of age or older
2. Self-reported daily smoker
3. Positive cotinine from urine sample
4. Motivated to quit smoking completely within five weeks of the Screening Visit (>5 on reported motivation)
5. Capable of and agree to complete study requirements
6. Literate in English, self-report
7. Must be available for the duration of study
8. Informed consent obtained

10. Must own study compatible smart-phone (iPhone or Android) 11. Must be a current resident of the United States

Exclusion Criteria for the Remote Cohort

1. Any self-report, diagnosis or treatment of heart attack, unstable angina, angioedema, seizures, cerebrovascular accident (CVA) within the last six months.
2. Any self-report, diagnosis or treatment of bipolar, schizophrenia or suicidal ideation within the last six months. (For suicidal ideation a score of ≥7 on the Suicidal Behavior Questionnaire, see Appendix 15)
3. Self-report of diagnosis or treatment for depression within the past six months, unless participant has written permission by their healthcare provider to participate
4. History of renal disease
5. Allergy to any of the ingredients in varenicline
6. Participation in another smoking cessation program or any type of clinical trial in the past 3 months
7. Use of any smoking cessation medication in the past three months
8. Any other medical condition(s) which the licensed study physician deems unacceptable for participation in this study
9. Consume greater than 21 alcohol drinks per week.
10. No two members of the same household may participate in this study
11. No study staff or their immediate family may participate in the study
12. Females who are pregnant, breast feeding, or not currently using a medically approved form of birth control and unwilling to do so.

Acceptable methods of birth control include abstinence, oral contraceptives, the contraceptive patch, the contraceptive ring, and condoms.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona State University, Phoenix, Arizona
  - Los Angeles Clinical Trials, Burbank, California

IPD SHARING:
Plan to Share IPD: Undecided
While the exact process is unclear, when all data have been locked and investigators have published what they choose, de-identified data will be made available for the duration that we are required by NIH to maintain the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1.0mg Varenicline b.i.d. | 0.5mg Varenicline b.i.d. | 0.0mg Placebo Varenicline b.i.d.
Started | 104 | 104 | 105
Completed | 70 | 66 | 76
Not Completed | 34 | 38 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.0mg Varenicline b.i.d. | 0.5mg Varenicline b.i.d. | 0.0mg Placebo Varenicline b.i.d. | Total
Number analyzed (Participants) | 104 | 104 | 105 | 313
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (10.5) | 51.4 (11.2) | 51.0 (12.3) | 51.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One person did not identify their sex, though we have all of the rest of their information. Thus, we actually have 104 participants in the 1.0 mg condition, but could only show 103 when reporting sex
  Participants
    number analyzed (Participants) | 103 | 104 | 105 | 312
    Female | 56 | 65 | 33 | 154
    Male | 47 | 39 | 72 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 60 | 58 | 63 | 181
  Race: African-American | 40 | 44 | 35 | 119
  Race: Asian | 0 | 1 | 2 | 3
  Race: AI/AN | 0 | 0 | 1 | 1
  Race: Other | 0 | 1 | 1 | 2
  Race: Missing | 4 | 0 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 104 | 104 | 105 | 313

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Have Continuous Abstinence as Verified by Breath Carbon Monoxide or Urine Cotinine
Description: Participants will provide self reported smoking status that has been verified by breath carbon monoxide or cotinine - Continuous abstinence
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1.0mg Varenicline b.i.d. | 0.5mg Varenicline b.i.d. | 0.0mg Placebo Varenicline b.i.d.
Number analyzed (Participants) | 104 | 104 | 105
Participants | 17 | 9 | 9

2. Secondary Outcome: Breath Carbon Monoxide or Urine Cotinine Verified Abstinence From Smoking Cigarettes - Point Prevalence Abstinence
Description: Participants will provide self reported smoking status that has been verified by breath carbon monoxide or cotinine - point prevalence abstinence
Time Frame: Week 12 visit
Measure: Count of Participants; unit: Participants
Arm/Group | 1.0mg Varenicline b.i.d. | 0.5mg Varenicline b.i.d. | 0.0mg Placebo Varenicline b.i.d.
Number analyzed (Participants) | 104 | 104 | 105
Participants | 25 | 12 | 9

3. Secondary Outcome: Breath Carbon Monoxide Verified Abstinence From Smoking Cigarettes
Description: Participants who self report not smoking will be asked to have smoking status verified by breath carbon monoxide
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | 1.0mg Varenicline b.i.d. | 0.5mg Varenicline b.i.d. | 0.0mg Placebo Varenicline b.i.d.
Number analyzed (Participants) | 104 | 104 | 105
Participants | 16 | 11 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were measured in relation to the baseline at weeks 2, 4, 8, 12, 13 and 26.
Description: No different
Arm/Group | 1.0mg Varenicline b.i.d. | 0.5mg Varenicline b.i.d. | 0.0mg Placebo Varenicline b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104 | 2/105
Other Adverse Events (participants affected / at risk) | 49/104 | 43/104 | 35/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0mg Varenicline b.i.d. (N=104) | 0.5mg Varenicline b.i.d. (N=104) | 0.0mg Placebo Varenicline b.i.d. (N=105)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stab Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Participant was stabbed in the community, and survived.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0mg Varenicline b.i.d. (N=104) | 0.5mg Varenicline b.i.d. (N=104) | 0.0mg Placebo Varenicline b.i.d. (N=105)
Nausea (Gastrointestinal disorders) | 30 (32) | 23 (23) | 8 (8)
Insomnia (General disorders) | 7 (7) | 3 (3) | 10 (10)
Irritability (Psychiatric disorders) | 6 (6) | 9 (9) | 10 (10)
Vivid Dreams (General disorders) | 22 (22) | 19 (19) | 17 (17)
Constipation (Gastrointestinal disorders) | 9 (9) | 9 (9) | 4 (4)

LIMITATIONS AND CAVEATS:
Note that the study was interrupted because of COVID.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT03557294/Prot_SAP_001.pdf